CLINICAL TRIAL: NCT05173831
Title: An Open-Label Feasibility and Safety Study of MDMA-Assisted Group Therapy for the Treatment of Posttraumatic Stress Disorder in Veterans
Brief Title: Study of Feasibility and Safety of MDMA-Assisted Group Therapy for the Treatment of PTSD in Veterans
Acronym: MPG1
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Transfer of Sponsorship
Sponsor: Lykos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MPG1
Record Dates: First submitted 2021-12-13; First posted 2021-12-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — N-Methyl-3,4-methylenedioxyamphetamine; Therapeutics

STUDY DESIGN:
Intervention Model Description: Open-label study examining safety and effects of two sessions of MDMA-assisted therapy each followed by four integrative therapy sessions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Two Sessions of MDMA-assisted therapy (Experimental): Two MDMA-assisted Therapy Sessions with 120 mg midomafetamine HCl and optional supplemental dose of 60 mg 1.5 to 2 hours later
  Interventions: Drug: Midomafetamine; Behavioral: Therapy

INTERVENTIONS:
Drug: Midomafetamine — Initial dose of 120 mg midomafetamine HCl and optional supplemental dose of 60 mg 1.5 to 2 hours later
  Other Names: 3,4-methylenedioxymethamphetamine; MDMA
Behavioral: Therapy — Manualized therapy performed by therapist team

SUMMARY:
The goal of this clinical trial is to learn if MDMA-assisted group therapy is safe and effective in in people with at least moderate PTSD.

The main question it aims to answer is: Do two sessions of open-label MDMA-assisted group therapy reduce PTSD symptoms?

Participants will undergo non-drug preparatory therapy sessions before their MDMA-assisted therapy sessions. After, they will undergo non-drug integrative therapy sessions.

DETAILED DESCRIPTION:
To further assess the feasibility and safety of MDMA-assisted group therapy for participants with at least moderate PTSD, the sponsor is conducting a Phase 2, open-label, non-randomized, 3-cohort study. This novel treatment package consists of two once-monthly Experimental Sessions of therapy combined with a divided-dose of MDMA (120 mg midomafetamine HCl and optional supplemental dose of 60 mg 1.5 to 2 hours later), along with non-drug preparatory and integrative therapy administered in both individual and group sessions.

The Primary Outcome measure, the Clinician Administered PTSD Scale (CAPS-5), evaluates changes in PTSD symptom severity and is assessed by a blinded centralized Independent Rater (IR) pool. The therapeutic approach will combine manualized MDMA-assisted therapy for PTSD with group therapy components.

ELIGIBILITY:
Inclusion Criteria:

* Are at least 18 years old.
* Are a U.S. Military Veteran
* Are fluent in speaking and reading the predominantly used or recognized language of the study site.
* Are able to swallow pills.
* Agree to have study visits recorded, including Experimental Sessions, outcome assessments, and non-drug psychotherapy sessions.
* Must provide a contact who is willing and able to be reached by the investigators in the event of a participant becoming suicidal or unreachable.
* Must agree to inform the investigators within 48 hours of any medical conditions and procedures.
* If able to become pregnant, must have a negative pregnancy test at study entry and prior to each Experimental Session, and must agree to use adequate contraception through 10 days after the last Experimental Session.
* Must not participate in any other interventional clinical trials during the duration of the study.
* Have a current PTSD diagnosis at the time of screening.

Exclusion Criteria:

* Are not able to give adequate informed consent.
* Have uncontrolled hypertension.
* Have a marked baseline QTcF interval >450 milliseconds [ms] demonstrated on repeated ECG assessments.
* Have a history of additional risk factors for Torsade de pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome).
* Have evidence or history of significant medical disorders.
* Have symptomatic liver or biliary disease.
* Have history of hyponatremia or hyperthermia.
* Weigh less than 48 kilograms (kg).
* Are pregnant or nursing, or are able to become pregnant and are not practicing an effective means of birth control.
* Have an active illicit drug or prescription drug substance use disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in CAPS-5 Total Severity Score | Baseline - 3 months from first Experimental Session
  The CAPS-5 is a semi-structured interview that assesses index history of DSM-5-defined traumatic event exposure [114], including the most distressing event, time since exposure, to produce a diagnostic score (presence vs. absence) and a PTSD Total Severity score [114]. The CAPS-5 rates intrusion symptoms (intrusive thoughts or memories), avoidance, cognitive and mood symptoms, arousal and reactivity symptoms, duration and degree of distress and dissociation. The total severity score is a sum of symptom frequency and intensity scores for the subscales B (re-experiencing), C (avoidance) and D (hypervigilance) and ranges from 0 to 136, with higher scores indicating greater severity of PTSD symptoms.

SECONDARY OUTCOMES:
Change in Sheehan Disability Scale (SDS) | Baseline - 3 months from First Experimental Session
  Sheehan Disability Scale (SDS) total score, a measure of clinician-rated functional impairment. The first three items indicate degree of impairment in the domains of work/school, social life, and home life, with response options based on an eleven-point scale (0=not at all to 10=extremely), and five verbal tags (not at all, mildly, moderately, markedly, extremely). The remaining two items assess Days Lost and Days Unproductive during the reporting period.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Stauffer, MD, Principal Investigator — Associate Professor of Psychiatry at Oregon Health & Science University